CLINICAL TRIAL: NCT02599506
Title: Fear of Cancer Recurrence (FoR) Trajectory During Radiation Treatment and Follow-up Into Survivorship of 100 Breast Cancer patients-a Pilot Study
Brief Title: Fear of Cancer Recurrence (FoR) Trajectory During Radiation Treatment
Acronym: FORECAST
Status: Completed | Type: Observational
Sponsor: University of St Andrews (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Prof G Humphris, Professor of Health Psychology, University of St Andrews
Other Study IDs: 20l5MaySP529
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; fear of recurrence; longitudinal study; radiation therapy; emotional concerns; trajectory; psychological constructs; diary keeping
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer radiation therapy: Observation over a period of all treatment sessions for radiotherapy

SUMMARY:
This pilot study concentrates on studying the trajectory of breast cancer patient's fear of recurrence (FoR) over the course of radiation therapy. The aim is to collect repeated ratings of 100 breast cancer patient's FoR over the course of their treatment. It is hypothesized that cancer patient's FoR level will rise on nearing the termination of the in radiotherapy treatment, and radiotherapist-patient interaction modifies the development of patient's FoR.

DETAILED DESCRIPTION:
The aim of this pilot study is to examine the collection of FoR levels in a longitudinal design with 100 breast cancer patients receiving radiotherapy for their disease. In this study, an intensive longitudinal design will be employed (Bolger & Laurenceau, 2013). There will be two data collection types. First, will be self-reported questionnaires. Patients will complete questions including three sections: 1) demographic information (i.e. age, education, employment, marital/family status), 2) a 7-item FoR scale (ACCRE FCR) and 3) a 20-item Affect Schedule (PANAS) before first radiation treatment (T1). Throughout the period of treatment, a 3-item FoR questionnaire (ACCRE FCR 3 Items) will be designed as a daily diary to monitor patient's FoR level. Then, at the end of the radiotherapy treatment (T2), PANAS will be measured again. Finally, six-eight weeks after the end of the treatment (T3), all participants will be asked to complete the 7-items FCR questionnaire once again as well as a 5-item EuroQoL EQ-5D-3L scale by telephone.

The second data collection media is audiotape. The conversations between radiotherapist and patient in the weekly review appointment will be recorded and a behavioural coding system (VR-CoDES) will be used to analyse the interactions between patient and radiotherapist.

Data analysis will involve statistical analysis and qualitative methods. Statistical analyses will be conducted using Statistical Package for the Social Sciences (SPSS) Analytics software v.22, Analysis of MOment Structures (AMOS) v.22 and MPlus™ (SEM: Structural Equation Modelling). Initial analysis will plot individual and group average curves over the days that patients are treated. The analysis will develop a statistical model based upon SEM principles of growth curves. Each patient is expected to disclose increased fears of recurrence over the course of treatment. Latent curve modelling will be developed to test the relationship of FoR over the time course of the treatment.

As part of this pilot study the investigators wish to investigate the appropriateness of these models and to test the extent of growth of FoR to the outcome at 6-8 weeks follow up, using the FoR 7 item measure. Covariates will be introduced for control purposes and indicate initial level of negative affectivity (The Positive and Negative Affect Schedule - PANAS), age and initial level of disease severity. Alternative strategies of analysis are considered appropriate and may enable a parallel strategy. This would involve a simpler approach concentrating on the raw data. Linear modelling (multi-level) which will include estimation of linear slopes being used to predict FoR outcome.

Audio recordings of the consultation will be transcribed verbatim in order to investigate how the radiotherapist-patient communication affects the development of FoR.

ELIGIBILITY:
Inclusion Criteria:

* Female patient who are diagnosed with breast cancer, age 18+

Exclusion Criteria:

* Under 18 years old
* Male
* Known psychiatric illness
* Receiving palliative radiotherapy (non-curative)
* Unable to communicate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, 100 breast cancer patients receiving radiotherapy at the Edinburgh Cancer Centre will be recruited.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Fear of Recurrence Level-ACCRE FCR | 6-8 weeks after treatment
  The ACCRE FCR scale has been employed in a national study, it ranges from 4-20. A score of 10 is a significant level (60th percentile) considered appropriate for the patient to receive a brief intervention.

SECONDARY OUTCOMES:
The Positive and Negative Affect Schedule (PANAS) | 4 weeks following baseline visit
  The Positive and Negative Affect Schedule (PANAS) is a 20-item self-report measure of positive and negative affect. The PANAS has been shown to possess adequate psychometric properties in a large sample drawn from the general adult population, and the construct validity of the PANAS scales and the reliabilities of both scales were adequate, Cronbach's α were 0.89 for Positive Affectivity and 0.85 for Negative Affectivity (Crawford & Henry, 2004).
5 EQ-5D-3L | 6-8 weeks after treatment
  The EQ-5D-3L is a standardised instrument for use as a measure of health outcome and was developed by the EuroQol Research foundation. It consists of five questions relating to five dimensions of health; mobility, self-care, usual activities, pain and discomfort and anxiety and depression. The EQ-5D has well-established validity and reliability and has been used in many studies of patients with a variety of chronic conditions in many different countries (Schrag et al., 2000; Walters & Brazier, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Gerald M Humphris, PhD, Principal Investigator — University of St Andrews
Locations (1):
- NHS Lothian Edinburgh Cancer Centre, Edinburgh, United Kingdom

REFERENCES:
- [Result] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Result] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Result] Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res. 2005 Aug;14(6):1523-32. doi: 10.1007/s11136-004-7713-0. PMID 16110932
- [Derived] Popov V, Ellis-Robinson A, Humphris G. Modelling reassurances of clinicians with hidden Markov models. BMC Med Res Methodol. 2019 Jan 9;19(1):11. doi: 10.1186/s12874-018-0629-0. PMID 30626327
- [Derived] Yang Y, Cameron J, Bedi C, Humphris G. Fear of cancer recurrence trajectory during radiation treatment and follow-up into survivorship of patients with breast cancer. BMC Cancer. 2018 Oct 20;18(1):1002. doi: 10.1186/s12885-018-4908-2. PMID 30342495
- [Derived] Humphris G, Yang Y, Barracliffe L, Cameron J, Bedi C. Emotional talk of patients with breast cancer during review appointments with therapeutic radiographers: effects on fears of cancer recurrence. Support Care Cancer. 2019 Jun;27(6):2143-2151. doi: 10.1007/s00520-018-4484-7. Epub 2018 Oct 1. PMID 30276473